CLINICAL TRIAL: NCT00927758
Title: Pilot Study to Examine the Post-Dose Changes in Exhaled Nitric Oxide (eNO) Following Treatment With Fluticasone Propionate (FP)/Salmeterol (SAL) Combination Product Advair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-Sandoz-2009-PilotFP
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2014-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Sequence 1: Flu/Sal- 250mcg/50mcg ->100mcg/50mcg->500mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg
- Sequence 2: Flu/Sal- 500mcg/50mcg ->250mcg/50mcg->100mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg
- Sequence 3: Flu/Sal- 100mcg/50mcg ->250mcg/50mcg->500mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg
- Sequence 4: Flu/Sal- 250mcg/50mcg ->500mcg/50mcg->100mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg
- Sequence 5: Flu/Sal- 500mcg/50mcg ->100mcg/50mcg->250mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg
- Sequence 6: Flu/Sal- 100mcg/50mcg ->500mcg/50mcg->250mcg/50mcg (Active Comparator): Treatment cycle 1: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
  Treatement Cycle 2 : Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
  Treatment Cycle 3: Patient randomized to Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
  There were 14 days washout period between cycles.
  Interventions: Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol (Flu/Sal) : 100mcg/50mcg, 250mcg/50mcg,500mcg/50 mcg — fluticasone propionate/salmeterol diskus
  Other Names: Advair DISKUS

SUMMARY:
To examine the post-dose changes in exhaled Nitric Oxide (eNO) following treatment with inhaled Advair in subjects with chronic but stable asthma as defined in Global Initiative for Asthma (GINA) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* must be able to speak, read, and understand English
* exhaled Nitrous Oxide levels must be greater than or equal to 60 ppb at screening and greater than or equal to 55 ppb at Visits 2, 9, and 16
* must have history of at least 6 months of chronic, but stable asthma
* except for the presence of asthma, subjects must be in general good health

Exclusion Criteria:

* past or present history of experiencing allergic reaction to medications used in this study
* subjects must not be receiving ongoing regular treatment with inhaled corticosteroids
* subjects must not have ragweed allergy
* subjects must have no recent history of respiratory infections for at least 1 month prior to screening and until the end of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - CompleWare, Iowa City, Iowa
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Actual screened patients was 105. However, 22 eligible patients were randomized.
Period: Treatment Cycle 1 (Day 1 - Day 7)
Arm/Group | Sequence 1: Flu/Sal- 250mcg/50mcg ->100mcg/50mcg->500mcg/50mcg | Sequence 2: Flu/Sal- 500mcg/50mcg ->250mcg/50mcg->100mcg/50mcg | Sequence 3: Flu/Sal- 100mcg/50mcg ->250mcg/50mcg->500mcg/50mcg | Sequence 4: Flu/Sal- 250mcg/50mcg ->500mcg/50mcg->100mcg/50mcg | Sequence 5: Flu/Sal- 500mcg/50mcg ->100mcg/50mcg->250mcg/50mcg | Sequence 6: Flu/Sal- 100mcg/50mcg ->500mcg/50mcg->250mcg/50mcg
Started | 4 ("Started " indicates randomized as well as safety set.) | 4 | 4 | 3 | 3 | 4
Intent to Treat (ITT) | 4 | 4 | 4 | 2 | 3 | 3
Completed | 4 | 4 | 4 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Period: Treatment Cycle 2 (Day 1 - Day 7)
Arm/Group | Sequence 1: Flu/Sal- 250mcg/50mcg ->100mcg/50mcg->500mcg/50mcg | Sequence 2: Flu/Sal- 500mcg/50mcg ->250mcg/50mcg->100mcg/50mcg | Sequence 3: Flu/Sal- 100mcg/50mcg ->250mcg/50mcg->500mcg/50mcg | Sequence 4: Flu/Sal- 250mcg/50mcg ->500mcg/50mcg->100mcg/50mcg | Sequence 5: Flu/Sal- 500mcg/50mcg ->100mcg/50mcg->250mcg/50mcg | Sequence 6: Flu/Sal- 100mcg/50mcg ->500mcg/50mcg->250mcg/50mcg
Started | 4 | 4 | 4 | 2 | 3 | 3
Per Protocol Population (PP) | 4 | 4 | 3 | 1 | 3 | 2
Completed | 4 | 4 | 3 | 1 | 3 | 2
Not Completed | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Did not meet eNO criteria | 0 | 0 | 1 | 1 | 0 | 1
Period: Treatment Cycle 3 (Day 1 - Day 7)
Arm/Group | Sequence 1: Flu/Sal- 250mcg/50mcg ->100mcg/50mcg->500mcg/50mcg | Sequence 2: Flu/Sal- 500mcg/50mcg ->250mcg/50mcg->100mcg/50mcg | Sequence 3: Flu/Sal- 100mcg/50mcg ->250mcg/50mcg->500mcg/50mcg | Sequence 4: Flu/Sal- 250mcg/50mcg ->500mcg/50mcg->100mcg/50mcg | Sequence 5: Flu/Sal- 500mcg/50mcg ->100mcg/50mcg->250mcg/50mcg | Sequence 6: Flu/Sal- 100mcg/50mcg ->500mcg/50mcg->250mcg/50mcg
Started | 4 | 4 | 3 | 1 | 3 | 2
Completed | 4 | 4 | 3 | 1 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Patients: Baseline measured for all randomized (safety set) patients.
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.86 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline (for Each Treatment Cycle) in Exhaled Nitric Oxide (eNO)
Description: Percentage change in eNO was reported following treatment with inhaled Advair in subjects with chronic but stable asthma as defined in Global Initiative for Asthma (GINA) guidelines. eNO was calculated 3 times every day in a treatment cycle for 7 days. The maximum value of all 3 collected value were collected for each seven days of the individual treatment cycle. Out of the maximum values, the minimum was taken and used for calculating the percentage change from baseline.
Time Frame: Baseline to Day 7 of each treatment cycle (total duration about 8 - 10 weeks)
Population: The per-protocol (PP) population was all subjects who completed the study with no major variances that would impair the analysis of the data
Measure: Mean (Standard Deviation); unit: Percentage change in eNO
Groups:
- Flu/Sal- 100mcg/50mcg: All randomized patients Fluticasone Propionate/Salmeterol (Flu/Sal) received 100mcg/50mcg once daily for 7 days.
- Flu/Sal- 250mcg/50mcg: All randomized patients Fluticasone Propionate/Salmeterol (Flu/Sal) received 250mcg/50mcg once daily for 7 days.
- Flu/Sal- 500mcg/50mcg: All randomized patients Fluticasone Propionate/Salmeterol (Flu/Sal) received 500mcg/50mcg once daily for 7 days.
Arm/Group | Flu/Sal- 100mcg/50mcg | Flu/Sal- 250mcg/50mcg | Flu/Sal- 500mcg/50mcg
Number analyzed (Participants) | 17 | 17 | 17
Percentage change in eNO | 36.65 (18.74) | 45.31 (16.46) | 54.58 (12.55)

ADVERSE EVENTS:
Description: Safety set includes all subjects who received at least one dose of drug.
Arm/Group | Flu/Sal- 100mcg/50mcg | Flu/Sal- 250mcg/50mcg | Flu/Sal- 500mcg/50mcg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 1/17
Other Adverse Events (participants affected / at risk) | 3/20 | 1/19 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flu/Sal- 100mcg/50mcg (N=20) | Flu/Sal- 250mcg/50mcg (N=19) | Flu/Sal- 500mcg/50mcg (N=17)
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flu/Sal- 100mcg/50mcg (N=20) | Flu/Sal- 250mcg/50mcg (N=19) | Flu/Sal- 500mcg/50mcg (N=17)
Viral Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Upper Respiratory infection (Infections and infestations) | 1 | 0 | 3
Worsening Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dilated, Dry Eyes (Eye disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Sandoz's agreements with its investigators may vary. However, Sandoz does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.